CLINICAL TRIAL: NCT03623425
Title: Comparison of PET Imaging With 68GA-PSMA-11 and 18F-Fluorocholine for the Identification of Site of Recurrence in Men With Prostate Cancer
Brief Title: Comparison of PET With 68GA-PSMA-11 and 18F-Fluorocholine for Recurrence in Men With Prostate Cancer
Acronym: TEPGALCHOL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: GIE NANCYCLOTEP (Other); Advanced Nuclear Medicine Ingredients (ANMI) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-003620-69; PSS2017/ANMI-OLIVIER/VS (Other: sponsor code)
Record Dates: First submitted 2018-08-06; First posted 2018-08-09 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Phase III, open, single center, prospective, controlled and randomized crossover study comparing diagnostic performance of 68GA-PSMA-11 and 18F-Fluorocholine. 68GA-PSMA-11 PET and 18F-Fluorocholine PET interpretation will be done by different nuclear physicians.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 68Ga-PSMA-11 PET before 18F-FCH PET (Experimental): Crossover design
  Interventions: Drug: 68Ga-PSMA-11 PET; Drug: 18F-FCH PET
- 18F-FCH PET before 68Ga-PSMA-11 PET (Experimental): Crossover design
  Interventions: Drug: 68Ga-PSMA-11 PET; Drug: 18F-FCH PET

INTERVENTIONS:
Drug: 68Ga-PSMA-11 PET — a 68GA-PSMA-11 PET exam before the a 18F-FCH PET exam
Drug: 18F-FCH PET — a 18F-FCH PET exam before the 68Ga-PSMA-11 PET exam

SUMMARY:
As choline transport and phosphorylation are upregulated in most cancers, including prostate cancer, positron emission tomography (PET) with choline tracers has found widespread use to detect recurrent disease. However, choline metabolism is not increased in a significant number of cases, probably explaining why this imaging method has been reported to be weakly sensitive and specific fro the detection of prostate cancer lesions, especially at low prostate-specific antigen (PSA) levels. By contrast, prostate-specific membrane antigen (PSMA) is overexpressed in most prostate cancer, suggesting that 68Ga-labelled PSMA ligands could be superior to choline tracers. A meta-analysis published in 2016 (Perera M. and al.), which included 18 studies, of which five reported histolopathologic correlation data for 68Ga-PSMA PET-positive lesions, indicated favourable sensitivity and specificity profiles of 68Ga-labelled PSMA ligands compared to choline-based PET imaging techniques.

DETAILED DESCRIPTION:
HBED-PSMA Sterile Cold Kit is a kit for preparation of radiolabelled 68Ga-PSMA-11. After radiolabelling with a 68Ga chloride solution complying with the requirements of monograph 2464 of the European Pharmacopoeia (Ph Eur), the solution may be used in men with biochemical relapse of prostate cancer after treatment. A large number of studies have been published on 68Ga-PSMA-ligands but none has yet been conducted with a product manufactured in accordance with ANMI technology. The aim of the study is to demonstrate the superiority of 68Ga-PSMA-11, prepared from a room temperature radiolabel kit containing PSMA-11 (PSMA-11 Sterile Cold Kit) and gallium 68 obtained from a 68Ge / 68Ga generator on 18F-Fluorocholine (18F-FCH) in identifying prostate cancer recurrence after radical treatment sites. So, patients will be evaluated with the current workup at CHRU of Nancy and will then be submitted to 68GA-PSMA-11 and 18F-FCH imaging. Patients will be randomized to the imaging procedure after workup in a 1/1 ratio between 68GA-PSMA-11 and comparator. So all patients will be submitted to 68GA-PSMA-11 and 18F-FCH; 50% of patients will receive the 68GA-PSMA-11 first; 50% of patients will receive the comparator first. There will be a time interval of minimum 7 days and maximum 14 days between both imaging procedures.

In order to mimic, as far as possible, the routine clinical practices, a sequential unblinding will be used for image readers. Readers will evaluate 68GA-PSMA-11 and 18F-FCH images with progressive access to more clinical information on each read. It will be done in three steps: fully blinded image evaluation, then image evaluation with results of the patient's clinical history and finally image evaluation with results of the patient's workup and clinical history.

ELIGIBILITY:
Inclusion Criteria:

* Adult men ranging in age from 18 to 80
* Patient who have developed prostate cancer, and underwent radical treatment by prostatectomy or radiotherapy.
* PSA<10 ng/ml at inclusion
* Rising prostate-specific antigen (PSA) after curative treatment of prostate cancer (radical prostatectomy or radiation therapy). Following definitions will apply:

  * Biochemical recurrence =

    * After surgery: two sequential PSA values >0.2 ng/ml
    * After radiation therapy: PSA increased by 2 ng/ml above nadir value
  * Residual disease =

    * After surgery: positive PSA immediately after surgery or positive surgical margin
    * After radiation therapy: two sequential PSA >0.2 ng/ml (to avoid false positive)
  * Progressive disease =

    * PSA doubling time ≤ 6 months irrespective of initial PSA value
* Patients with a positron emission tomography with 18F-Fluorocholine (PET 18F-Fcholine) requested, as part of routine care.
* Estimated life-expectancy > 6 months
* Patients able to come for PET exams
* Patients affiliated to or beneficiary of a social security plan
* Patients physically and psychologically able to participate to the study
* Person informed about study organization and having signed the informed consent
* Patients who understood the principle and modalities of the study
* Person undergone the medical examination adapted to research

Exclusion Criteria:

* Known hypersensitivity to the active substance or to any excipient of the IMP
* Patients with known allergy to furosemide or sulfonamides. Other contraindications to furosemide do not apply to patients for whom the product will be used as a single dose
* Patients with a history of malignant pathology (except for basal-cell cutaneous carcinoma)
* Drug or alcohol dependence, serious current illness, mental disorder or any circumstance which, in the opinion of the investigator, could interfere with the conduct or interpretation of the study
* Exposure to another IMP within 60 days prior to inclusion
* Person referred in articles L.1121-7 and L.1121-8 of the Public Health Code:

  * Minor person (non-emancipated)
  * Adult person under legal protection (any form of public guardianship)
  * Adult person incapable of giving consent
* Person deprived of liberty for judicial or administrative decision, Person under psychiatric care according to articles L. 3212-1 and L. 3213-1.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer is an only men disease
Enrollment: 46 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Number of lesions characteristic for prostate cancer detected by each TEP imaging method, by 68Ga-PSMA-11 and 18F-Fluorocholine | three months after the last PET exam for each patient
  An experts committee will conduct a confirmatory assessment of all lesions three months after the last PET scan for each patient..

SECONDARY OUTCOMES:
Count and characterize prostate cancer lesions for each method | three months after the last PET exam for each patient
  Detection rate and Standardized Uptake Value (SUV) and tumor to background ratio (TBR)
Number of patients whose diagnosis and/or treatment are impacted by the results of the imaging procedures | three months after the last PET exam for each patient
  Compare diagnoses and treatments decided with and without PET results
Sensitivity, specificity and predictive values of each tomography method | three months after the last PET exam for each patient
  + 95% CI
Number of adverse events and serious adverse events, whether or not related to research | three months after the last PET exam for each patient
  Description of adverse events, incidence, severity, outcome and causality

CONTACTS AND LOCATIONS:
Overall Officials: Pierre OLIVIER, MD, PhD, Principal Investigator — CHRU de NANCY- BRABOIS
Locations (1):
- CHRU de NANCY- BRABOIS, Vandœuvre-lès-Nancy, France